CLINICAL TRIAL: NCT05678790
Title: The Effect of 6-week Rehabilitation Program in Brothers With MPAN: A Report of Two Cases.
Brief Title: Mitochondrial Membrane Protein Neurodegeneration (MPAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Ömer Faruk ÖZÇELEP, Researcher, Kirsehir Ahi Evran Universitesi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEvran
Record Dates: First submitted 2022-12-22; First posted 2023-01-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: MPAN
Keywords: MPAN; Exercise Therapy; Balance and Coordination
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Case Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Balance and Coordination (Experimental): Since it is a case study, there will be only one group in the study.
  Interventions: Other: Passive Stretching; Other: Mobilization; Other: Muscle strengthening; Other: Balance and Coordination

INTERVENTIONS:
Other: Passive Stretching — Sustained passive stretching of hamstring, tendo-achilles, and adductors 10 (30 s, with three repetitions, five times per week)
Other: Mobilization — Grade four mobilizations is a stretching motion performed at the talocrural joint with anterior-posterior gliding. Mobilization was performed once a day, 6 times a day, and 5 times a week, only on both deformed feet of the older sibling
Other: Muscle strengthening — Abdominal muscle strengthening exercises were given to both siblings once a day, 10 times a day, 5 times a week. In the supine position, the patients were asked to lie on their knees with the knees flexed. The hip extensors were trained in the prone position on the bed by resisting hip extension
Other: Balance and Coordination — The following exercises were applied 5 times a week, with 1o repetition once a day.
  * Standing on one leg in front of the mirror,
  * Tandem walking,
  * Rhythmic Dynamic Stabilization,
  * Swiss ball sitting (eyes open and closed),
  * Counting the alphabet or numbers while marching

SUMMARY:
The purpose of this case study was to investigate the effects of therapeutic intervention in 9- and 12-year-old brothers with MPAN. The main hypothesis it aims to answer is:

-A 6-week balance and coordination focused rehabilitation program improves independence and gait parameters in patients with MPAN.

DETAILED DESCRIPTION:
Neurodegeneration with brain iron accumulation (NBIA) comprises a heterogeneous group of disorders with accumulation of iron in the brain, mostly basal ganglia. Mutations within C19orf12 have recently been identified in patients with NBIA. This C19orf12 gene -located in mitochondria and endoplasmic reticulum- encodes a mitochondrial membrane protein and the abbreviation MPAN. Pathogenic mutations in this gene are postulated to cause dysfunction of lipid homeostasis in mitochondria.

Patients with MPAN typically present with gait disturbance due to lower limb spasticity and dystonia, parkinsonism with subsequent spastic paresis, dysarthria, cerebellar ataxia, behavioral problems, dementia, psychomotor delay, peripheral neuropathy, visual changes like optic atrophy as well as bowel/bladder incontinence; however, MPAN has a greater variability compared with other NBIA cases in terms of age of onset (age three to 30 years) and speed of progression.

This study aims to investigate the effects of therapeutic intervention in male brothers, age 9 and 12, with MPAN. In particular, this study tested the following hypotheses after 6 weeks of rehabilitation by measuring muscle strength, muscle tone, range of motion , balance and coordination: (1) After the training period, muscle strenght, muscle tone and range of motion would be improved, (2) these developments in body function can lead to increase balance and coordination, and (3) due to the these improvements, functional independency may increase.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with MPAN

Exclusion Criteria:

* being involved in any other rehabilitation program

Ages: 9 Years to 14 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Balance | 6 weeks
  Balance and coordination will be evaluated with the Pediatric Berg Balance Test.
Functional İndependence | 6 weeks
  Functional independence which will evaluate with Functional Independence Measure for Children (WeeFIM).
Observational Gait Analysis | 6 weeks
  Gait characteristic will assessed with Observational Gait Analysis (OGA).

CONTACTS AND LOCATIONS:
Overall Officials: Figen TUNCAY, Study Director — Kirsehir Ahi Evran Universitesi
Locations (1):
- Ahi Evran University, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared online if requested.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months study finished

REFERENCES:
- [Background] Ramesh R, Deenadayalu A, Bhattacharjee S, Paramanandam V. C19orf12 mutation causing mitochondrial membrane-protein Associated Neurodegeneration masquerading as spastic paraplegia. Parkinsonism Relat Disord. 2021 Aug;89:146-147. doi: 10.1016/j.parkreldis.2021.07.014. Epub 2021 Jul 13. PMID 34298215
- [Background] Yang Y, Zhang S, Yang W, Wei T, Hao W, Cheng T, Wang J, Dong W, Qian N. Case Report: Identification of a De novo C19orf12 Variant in a Patient With Mitochondrial Membrane Protein-Associated Neurodegeneration. Front Genet. 2022 Mar 30;13:852374. doi: 10.3389/fgene.2022.852374. eCollection 2022. PMID 35432442